CLINICAL TRIAL: NCT03457675
Title: Development of Adaptive Deep Brain Stimulation (aDBS) for the Treatment of Intractable OCD: Phase Ia Using Activa PC+S
Brief Title: Development of Adaptive Deep Brain Stimulation for OCD (Phase 1a)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Pittsburgh (Other); Brown University (Other); Carnegie Mellon University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Principal Investigator, Wayne Goodman MD, Principal Investigator, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H40255; 1UH3NS100549 (NIH); 49340 (Other Grant/Funding Number: BCM ID)
Record Dates: First submitted 2017-08-14; First posted 2018-03-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep Brain Stimulation (DBS); Treatment Resistant OCD; Intractable OCD; Obsessive Compulsive Disorder (OCD); Cognitive Behavior Therapy (CBT); Exposure and Response Prevention (ERP)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: At the end of month 8 after DBS implant, all subjects will enter a one-month delayed onset withdrawal period in which the subject and Independent Evaluators are blinded to timing of discontinuation. See description below.
Who Masked: Participant, Outcomes Assessor
Masking Description: In all cases, the sequence will be as follows in one-week segments: 100% Active, 50% Active, Sham and Sham. Subjects will be seen weekly. Amplitude will be reduced by 50% at start of week 2 and turned off at start of week 3. Subjects will be told that DBS will be discontinued at some point during the 4 weeks. The purpose of the 50% initial reduction is to minimize rebound effects. The programmer (not the PI in this case) will be open to the design and perform "sham" activation. Relapse is defined as a 25% increase of the Y-BOCS over two consecutive visits compared to discontinuation baseline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Activa PC+S DBS implant for OCD (Experimental): all subjects will receive surgical implantation of DBS system
  Interventions: Device: Activa PC+S DBS implant for OCD
- One Month Blinded Discontinuation Period (Experimental): all subjects will enter a one-month blinded discontinuation period to confirm clinical benefit at the end of Month 8.
  Interventions: Other: One Month Blinded Discontinuation Period

INTERVENTIONS:
Device: Activa PC+S DBS implant for OCD — DBS system consists of the Activa PC+S Neurostimulation System:
  Model 37604 Activa PC+S Neurostimulator Model 37087 DBS Extension Model 37441 Patient Programmer Model 8181 Sensing Programmer Model 8180 Sensing Programmer Software Nexus D2/D3 System Nexus D2/D3 Application Programming Interface (API) Dow Corning Medical Adhesive, Medtronic Part #080118 Model 3387/3389 DBS Leads Model 37022 External Neurostimulator Model 8840 N'Vision Clinician Programmer Model 8870 Application Card Model 37642 Patient Programmer Model 37092 Patient Programmer Antenna
  Other Names: Deep Brain Stimulation System; DBS; Activa PC+S System
  Arms: Activa PC+S DBS implant for OCD
Other: One Month Blinded Discontinuation Period — The subject and Independent Evaluators are blinded to timing of discontinuation. In all cases, the sequence will be as follows in one-week segments: 100% Active, 50% Active, Sham and Sham. Subjects will be seen weekly. Amplitude will be reduced by 50% at start of week 2 and turned off at start of week 3. Subjects will be told that DBS will be discontinued at some point during the 4 weeks. The purpose of the 50% initial reduction is to minimize rebound effects. The programmer (not the PI in this case) will be open to the design and perform "sham" activation as described previously. Relapse is defined as a 25% increase of the Y-BOCS over two consecutive visits compared to discontinuation baseline.
  Arms: One Month Blinded Discontinuation Period

SUMMARY:
This research study is for participants that have been diagnosed with intractable Obsessive -compulsive disorder (OCD). OCD is a persistent and oftentimes disabling disorder marked by unwanted and distressing thoughts (obsessions) and irresistible repetitive behaviors. OCD affects 2-3% of the US population, and is responsible for substantial functional impairment and increased risk of early death.

The only established first-line treatments for OCD are cognitive-behavioral therapy (CBT) with exposure/response prevention and certain medications. About 30-40% of patients fail to respond and few experience complete symptom resolution. Up to 25% of patients have difficulty tolerating CBT and the risk of relapse after therapies remains large. For the most severe cases, neurosurgery (surgery in the brain), has long been the option of last resort.

In this study the investigators want develop an adaptive Deep Brain Stimulation (aDBS) system to use in subjects with intractable (hard to control) OCD. Deep brain stimulation remains investigational for OCD patients and is not considered standard therapy. DBS involves the surgical implantation of leads and electrodes into specific areas of the brain, which are thought to influence the disease. A pack implanted in the chest, called the neurotransmitter, keeps the electrical current coursing to the brain through a wire that connects the neurotransmitter and electrodes. It is believed deep brain stimulation may restore balance to dysfunctional brain circuitry implicated in OCD. The goal of this study is to enhance current approaches to DBS targeting in the brain and to use a novel approach to find a better and more reliable system for OCD treatment.

Phase Ia is to gather data to eventually develop a prototype adaptive DBS system for intractable OCD that uses signals from the brain to automatically adjust the DBS stimulation factors. The overall goal is to improve symptom management and reduce stimulation-induced behavioral side effects.

DETAILED DESCRIPTION:
RECRUITMENT:

Potential participants will be referred to our program by their treating clinicians, who will be made aware of our study through direct clinician-clinician letters and emails. Subjects may also learn of the study through consumer advocacy groups such as the International OCD Foundation (IOCDF), local non-profit organizations and local support group meetings and through the normals avenues that they share information.

ENROLLMENT:

A subject is considered enrolled upon signing informed consent, deemed eligible to be screened by the investigator. Decision-making capacity, which includes understanding, appreciation, reasoning and ability to express a choice, will be assessed as part of the informed consent process. The informed consent process will include discussions with the patient's family and referring clinician. Medical records will be carefully reviewed to determine adequacy of past treatments including CBT.

SCREENING:

Potential subjects meeting inclusion/exclusion criteria and willing to participate in the study as demonstrated by signing the informed consent will be enrolled in the study and undergo screening.

After the participant signs the required documents, he/she will undergo two baseline evaluations spaced over an approximate 1 month period. Diagnostic and screening ratings are completed, followed by complete medical, neurological and neurosurgical evaluations. The raters will be trained and certified in the use of the clinician-administered scales of the study. The purpose of the screening evaluations is to demonstrate that subject is in a stable clinical situation including a stable medical regimen, and are severely symptomatic. If this is the case, and they continue to meet inclusion/exclusion criteria, the participant will proceed to treatment (surgery to implant the DBS system. Final selection of candidates will be made by consensus of the multi-disciplinary investigator team ("Project Advisory Committee").

TREATMENT:

Subjects treated in Phase 1a will undergo a single stage DBS surgery, in which bilateral deep brain leads will be implanted under conscious sedation, followed by implantation of a single Implantable NeuroStimulator (INS), Activa PC+S, under general anesthesia.

1. A head CT will be performed on the morning of surgery for stereotactic planning.
2. Employing local anesthetic (with or without sedation as clinically indicated), a stereotactic headframe (Leksell Model G, Elekta Instruments, Atlanta, GA, USA) will be attached to the subject's skull on the morning of surgery in the operating room.
3. A 3D volumetric image (O-Arm 2, Medtronic Inc,, Boulder, CO, USA) will be performed for purposes of defining the volumetric stereotactic headspace.
4. The images will be uploaded onto a Computer Workstation (Stealth S7, Medtronic, Inc., Boulder, CO, USA) equipped with stereotactic planning software (Cranial 3.0) for the purpose of planning the surgery. The preoperative 3T MRI obtained prior to the surgical date, will be fused with the CT scan in the surgical planning station. The initial target point within the ventral striatum will be chosen based on the subject's specific anatomy. The surgical trajectory to this point will also be planned in order to avoid prominent vessels, the sulci, and the ventricles. The computer will generate the X, Y and Z coordinates to set on the frame as well as the coronal and sagittal angles of approach required to establish the desired trajectory and target point. This initial target point will be modified by the subject's specific anatomy as determined by the preoperative 3T MRI. The final target coordinates will be determined during this analysis.
5. While the surgeon is planning the procedure, the subject will be positioned supine on the operating table. A Foley catheter will be inserted. Antibiotics will be administered intravenously and vital signs will be monitored. The stereotactic head frame will be fixed to the operating table for subject safety, with the head elevated for subject comfort. A sterile prep and drape will be performed.
6. The target coordinates will be set on the stereotactic frame bringing the target point to the center of the operating arc. Additional local anesthetic will be given at the point of incision. Following incision, a 14 mm burr hole will be made employing a self-stopping perforator. The burr hole cap provided with the DBS lead will be secured to the skull with two screws. The dura will be coagulated and incised. The pial surface will be gently coagulated and a small incision will be made to allow easy entry of the electrode guides, which will be inserted to the brain according to standard stereotactic protocol.
7. A microelectrode (MER) probe will be inserted through the cannula and advanced in sub mm steps until the target is reached. Intraoperative image guidance will be obtained to ensure the MER probe is not mechanically deviated from target. If a deviation is identified, the stereotactic headframe will be adjusted accordingly.
8. Once the above adjustments have been made, the DBS quadripolar electrode (model 3387; Medtronic Inc., Minneapolis, MN, USA) will be inserted through the guide tube to the target point. Reticles will be attached to the frame and intraoperative imaging will be employed to confirm that the lead tip is positioned at the target and assess for the presence of intracerebral hemorrhage. Sedation will be withdrawn. An extension cable will be connected to the lead sterilely and the other end will be passed off the field to be connected to an external pulse generator so that test stimulation may be performed. Test stimulation will be performed via each contact to 1) assess for stimulation-induced side effects and 2) monitor for acute changes in behavior using a Likert-type scale to assess anxiety, arousal, and mood.
9. Intra-operative X-ray imaging may be performed as needed (up to 4 times per side) to ensure proper target has been reached.
10. A post-implantation 3D volumetric scan will be performed to confirm the electrode position.
11. Intra operative MER and behavioral testing of Stimulation with AFAR video recording will be performed.
12. Steps 5-9 above will be performed to insert the second electrode on the other side of the brain to complete implantation of both electrodes.
13. If there are no untenable side effects, the leads will be secured to the skull with the burr hole caps. The free end of the leads will be left in the sub-galeal space and the incisions will be closed in anatomical layers.
14. The headframe will be removed and general anesthesia will be induced. The Activa PC+S pulse generator will then be implanted and connected to the brain lead via extension cables.
15. A post-operative CT scan will be performed prior to discharge -to ensure that an intracerebral hemorrhage has not occurred.
16. The subject will be taken to the Recovery Room or the Neurosurgery ICU for post-operative monitoring (See below) and will be discharged from the hospital after at least one night of observation and when clinically stable. A Basic Metabolic Panel (BMP) may be run on the subject to confirm they are clinically stable.
17. The subject will return to the neurosurgery clinic (Visit 4) for post-operative evaluation according to normal clinical practice (approx 1 week after surgery). The wounds will be inspected and the subject's neurological status will be assessed. Sutures will be removed.

The subject will return to clinic about 2 weeks post-surgery for their post-surgical psychiatric symptom baseline and recording visit (Visit 5). Programming of the DBS device will occur at Visit 6, 1 week later.

The subject will return to clinic every 2 weeks for the first 2 months following the system activation. Each visit will last about 3-4 hours and will include clinician administered assessments, self-rated assessments, recordings and tasks to be performed.

Post-surgical 1.5 rs-fMRI scans will also be performed according to Medtronic standard post-implant MRI guidelines for deep brain stimulation systems to ensure safety.

Participants will be asked to keep their current medications constant for the first 6 months post-surgery. However, clinical circumstances which mandate changes will be allowed and notated should this occur.

Provocation Tasks:

The Provocation OC task (Provoc) and the Trier Social Stress Test (TSST) will be used to start OC-related distress and distress unrelated to OCD (e.g., performance anxiety), respectively. Three sessions will be videotaped with Automated Facial Affect Recognition (AFAR) system concurrent to recording of local field potentials (LFPs) from VS and scalp electroencephalography (EEG).

CBT Augmentation:

Starting at Month 7, subjects will receive a two-month (15 session) cognitive behavioral therapy (CBT) course where exposure and response prevention (ERP) for OCD will be delivered. Subjects already receiving stable CBT will be allowed to continue it during the study. Instead, we have developed standardized instructions to encourage exposure and resist compulsions (ERP) during this portion of the trial. Participants will be encouraged at study visits to actively confront OC triggers while refraining from ritual engagement. Subjects, especially those who are still habitually avoiding, will be given the opportunity to derive maximal clinical benefit by receiving a two-month "refresher" course of CBT prior to entering the double-blind discontinuation phase at 9 months.

Double Blinded Discontinuation:

The purpose of the one-month blinded discontinuation period is to confirm clinical benefit. At the end of month 8, subjects will enter a one-month delayed onset withdrawal period in which the subject and Independent Evaluators are blinded to timing of discontinuation. The decision whether to reinstate active DBS at the end of the discontinuation will be based on clinical considerations in discussion with the subject and significant others. The benefits and discomforts will be carefully weighed in arriving at a long-term plan. Escape criteria will include withdrawing consent or significant clinical deterioration warranting unblinding or reinstatement of treatment. Following exit from the discontinuation period, treatment will recommence as clinically indicated, including stimulation resumption or continued observation with the device off.

Monthly Programming/Classification/Evaluation Visits until End of Study (EOS):

Months 10-18 (Visits 20-28) - Following exit from the discontinuation phase based on clinical indication, treatment will recommence as clinically indicated around Month 10, including stimulation resumption or continued observation with device off. Refining state classifications and testing machine learning will continue, if stimulation is reinstated. Subjects that participated in the discontinuation phase will be considered off-treatment once Month 18 visit (Visit 298) has occurred.These visits will take place monthly for 9 months. Each visit will last approximately 3-4 hours.

Long-Term Follow-Up:

After the 18 months of the study, the device will remain implanted in those subjects who are doing well clinically. For subjects who are not responsive, it will be explanted, if the surgical risks of explantation are deemed acceptable by the treatment team. The follow-up management will be arranged on a case-by-case basis, depending on geographic location and desires of the subject, and DBS therapy management by our team will be guaranteed for at least two years if subjects continue to receive DBS therapy and do not arrange alternative management during that period. Attempts will be made to collect all device-related adverse events in all willing participants at 6-month intervals after they exit the currently proposed study.

Subject participation is anticipated to continue for a minimum of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* OCD DBS Subject Inclusion criteria:

  1. Signed informed consent prior to any study specific procedures being performed
  2. Male or female between ages 21 and 70;
  3. At least a five-year history of treatment-refractory OCD that causes substantial subjective distress and impairment in functioning;
  4. Y-BOCS minimum score of 28;
  5. Failed an adequate trial of at least three of the following SSRIs:

     Fluoxetine; fluvoxamine; citalopram; escitalopram; sertraline; paroxetine;
  6. Failed an adequate trial of clomipramine;
  7. Failed augmentation of one or more of the aforementioned drugs with at least one of the following antipsychotics: haloperidol; risperidone; quetiapine; ziprasidone; aripiprazole;
  8. Failed an adequate trial of CBT for OCD, defined as 25 hours of documented exposure and response prevention (ERP) by an expert therapist;
  9. Stable psychotropic medical regimen for the month preceding surgery
* Non-Implanted Control Subject Inclusion criteria:

  1. Signed informed consent prior to any study specific procedures being performed
  2. Male or female between ages 21 and 70
* Implanted ET Subject Inclusion criteria:

  1. Signed informed consent prior to any study specific procedures being performed
  2. Male or female between ages 21 and 70
  3. Diagnosed with Essential Tremor (ET) chronically, EXCLUDING head tremor, and implanted with DBS

Exclusion Criteria:

* OCD DBS Subject Exclusion criteria:

  1. Inability or refusal to give informed consent.
  2. Lifetime diagnosis of psychotic disorders such as schizophrenia;
  3. Alcohol or substance abuse/dependence within 6 months, excluding nicotine;
  4. Deemed at high risk of suicidal behavior or impulsivity, per clinical opinion assessments.
  5. Any Neurological/Medical condition that makes the subject, in the opinion of the surgeon, a poor candidate.
  6. Pregnant (confirmed by serum pregnancy test on females of child bearing age) or plans to become pregnant in the next 24 months.
  7. Need for Diathermy
  8. Contraindications to MRI
* Non-Implanted Control Subject Exclusion criteria:

  1. Inability or refusal to give informed consent.
  2. Lifetime diagnosis of mental illness
  3. A score of 8 or greater on part B of the Florida Obsessive Compulsive Inventory
  4. Any neurological disorders (i.e., MS, Parkinson's Disease, seizure disorders, etc.) or evidence of brain abnormalities/injury, such as tumor, stroke, or traumatic brain injury
  5. Pregnant (confirmed by self-report for females of child bearing age)
  6. Contraindications to MRI
* Implanted ET Subject Exclusion criteria

  1. ET subjects (with DBS implanted), WITH head tremor, may exacerbate artifact, therefore they will be excluded.
  2. Inability or refusal to give informed consent.
  3. Lifetime diagnosis of mental illness
  4. A score of 8 or greater on part B of the Florida Obsessive Compulsive Inventory
  5. Any other neurological disorder other than ET (i.e., MS, Parkinson's Disease, seizure disorders, etc.) or evidence of brain abnormalities/injury, such as tumor, stroke, or traumatic brain injury
  6. Contraindications to MRI

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects that display biomarkers of OCD-related distress | Month 6
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of OCD-related distress | Month 9
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of OCD-related distress | Month 12
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of OCD-related distress | Month 18
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with OCD-related distress during task exposure in clinic.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 6
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 9
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 12
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.
Percent of subjects that display biomarkers of DBS-induced hypomania | Month 18
  electrophysiological signals (deep brain local field potentials with scalp electroencephalography) from the brain showing Cohen's kappa k > 0.40, chance corrected classification agreement with DBS therapy during clinical visits.

SECONDARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Rating OCD Symptom Severity | Baseline to 30 days
  measured after closed-loop stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Goodman, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided